CLINICAL TRIAL: NCT06232772
Title: Research on Novel Biomarkers for Early Diagnosis of Parkinson's Disease:An Observational, Multicenter, Non-Randomized Controlled Study
Status: Recruiting | Type: Observational
Sponsor: Yousheng Xiao (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangxi University of Traditional Chinese Medicine (Unknown); Guilin Medical College (Other); Guangxi International Zhuang Medical Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Yousheng Xiao, professor, Guangxi Medical University
Organization: Guangxi Medical University (Other)
Other Study IDs: YXiao
Record Dates: First submitted 2024-01-20; First posted 2024-01-31 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- patients with clinically defined PD: Using an ELISA kit and α- Synuclein Ultrafine Fluorescence Detection Method to analyze the skin and body fluids of the included subjects α- synuclein level detection.
  Interventions: Diagnostic Test: α- Synuclein Ultrafine Fluorescence Detection Method
- patients with clinically probable PD: Using an ELISA kit and α- Synuclein Ultrafine Fluorescence Detection Method to analyze the skin and body fluids of the included subjects α- synuclein level detection.
  Interventions: Diagnostic Test: α- Synuclein Ultrafine Fluorescence Detection Method
- MSA group: Using an ELISA kit and α- Synuclein Ultrafine Fluorescence Detection Method to analyze the skin and body fluids of the included subjects α- synuclein level detection.
  Interventions: Diagnostic Test: α- Synuclein Ultrafine Fluorescence Detection Method
- PSP group: Using an ELISA kit and α- Synuclein Ultrafine Fluorescence Detection Method to analyze the skin and body fluids of the included subjects α- synuclein level detection.
  Interventions: Diagnostic Test: α- Synuclein Ultrafine Fluorescence Detection Method
- healthy subjects of equal age and sex without any risk or prodromal factor for PD: control group Using an ELISA kit and α- Synuclein Ultrafine Fluorescence Detection Method to analyze the skin and body fluids of the included subjects α- synuclein level detection.
  Interventions: Diagnostic Test: α- Synuclein Ultrafine Fluorescence Detection Method

INTERVENTIONS:
Diagnostic Test: α- Synuclein Ultrafine Fluorescence Detection Method — This technology belongs to the detection of a-syn aggregates in extracranial tissues, which can replace brain biopsy operations that are difficult to carry out clinically, thus breaking through the limitations of clinical experience in diagnosing a-synuclein lineage diseases and greatly improving the diagnostic and differential diagnostic level of this group of diseases.

SUMMARY:
This observational, multicenter, non-randomized controlled study is to evaluate the detection ability of α-Synuclein Ultrafine Fluorescence Detection Method for body fluids (Such as saliva, urine, cerebrospinal fluid, and blood, etc.) and skin in Parkinson's patients.

DETAILED DESCRIPTION:
Social benefits: This technology has minimal harm (skin sampling diameter of 1mm), rather than surgical traumatic brain biopsy, which meets the minimum harm and maximum benefit; 1) Clear clinical diagnosis and differential diagnosis of diseases at once, avoiding repetitive examinations, effectively saving medical expenses and medical insurance funds; 2) Beneficial for early diagnosis and intervention, reducing social and economic burden; 3) Enhance the disease diagnosis and treatment capabilities of the region, enhance basic medical research, and enhance the medical level of the region. Clinical advantage: This technology belongs to extracranial tissues α-Syn aggregate testing can replace brain biopsy procedures that are difficult to carry out clinically, thus breaking through the limitations of clinical experience in diagnosing a-synuclein lineage diseases and greatly improving the diagnostic and differential diagnostic level of this group of diseases.

Clinical needs: α-Synaptic nucleoprotein lineage diseases (Parkinson's disease, multisystem atrophy, and Lewy body dementia) have complex early symptoms, making diagnosis and differential diagnosis difficult. Early diagnosis is crucial for disease prognosis. Authoritative theories suggest that brain tissue biopsy is necessary for the diagnosis of this group of diseases, but it is difficult to generalize in clinical practice. Therefore, there is a 20% misdiagnosis and missed diagnosis rate in the clinical diagnosis of α-synaptic nuclear protein spectrum diseases. The α-Synuclein Ultrafine Fluorescence Detection Method for body fluids and skin in Parkinson's patients can truly reflect the degree of pathological aggregation in synapses, which is helpful for early diagnosis and evaluation of diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically defined or probable PD：According to the 2015 MDS diagnostic criteria, patients diagnosed with "clinically confirmed PD" regardless of age, gender, and meeting Hoehn&Yahr staging ≤ 2.5 were included as case group one, which met [Parkinson's syndrome+at least two supportive criteria+no absolute exclusion criteria]
* Patients with clinically probable PD：According to the 2015 MDS diagnostic criteria, patients diagnosed with "clinically probable PD", regardless of age or gender, and meeting Hoehn&Yahr staging ≤ 2.5 were included as case group two, i.e. patients who met [Parkinson's syndrome+no absolute exclusion criteria+1/2 supportive criteria+1/2 warning signs]
* MSA group：Adult onset (>30 years old), sporadic and progressive development, and possessing the following characteristics: 1 Has one of the following two conditions: ① Parkinson's syndrome with levodopa adverse response (bradykinesia, accompanied by muscle rigidity, tremors, or postural instability), ② cerebellar dysfunction: gait ataxia, accompanied by cerebellar articulation disorders, limb ataxia, or cerebellar eye movement disorders; 2. At least one manifestation of autonomic dysfunction is present: ① urinary incontinence (inability to control bladder urination, male with erectile dysfunction), ② orthostatic hypotension (a decrease in systolic blood pressure of ≥ 30mmHg and/or diastolic blood pressure of ≥ 15mmHg after standing for 3 minutes).
* PSP group：Clinical diagnosis and likely PSP included in the Chinese progressive supranuclear palsy clinical diagnostic criteria developed by the Parkinson's disease and motor disorders group of the Neurology Branch of the Chinese Medical Association in 2016;
* Healthy subjects：Healthy population matched with age and gender in the experimental group In addition to the selected patients, a study will also be conducted on patient data in the reference database of the proposing institution.

Exclusion Criteria:

* Patients who do not consent to study participation
* Secondary Parkinson's syndrome caused by vascular factors, drugs, etc
* Severe cognitive impairment, AD, amyotrophic lateral sclerosis and other neurodegenerative diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1) patients with clinically defined PD; 2) patients with clinically probable PD; 3) MSA group; 4) PSP group; 5) healthy subjects of equal age and sex without any risk or prodromal factor for PD.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1（Accuracy and precision） | 3 years
  To define test accuracy and precision of skin biopsy and body fluid detection of α-Synuclein Ultra Fine Fluorescence Method.
Primary Outcome 2（Sensitivity and specificity） | 3 years
  To define sensitivity and specificity of skin biopsy and body fluid detection of α-Synuclein Ultra Fine Fluorescence Method.

CONTACTS AND LOCATIONS:
Overall Officials: Yousheng Xiao, Professor, Principal Investigator — Guangxi Medical University
Locations (1):
- Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided